CLINICAL TRIAL: NCT06364306
Title: oPen Versus RobotIc retrOmuscular Repair in Medium to Large Ventral Hernias - the PRIOR Multicentre Randomized Controlled Trial
Brief Title: oPen Versus RobotIc retrOmuscular Repair in Medium to Large Ventral Hernias
Acronym: PRIOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: St. Clara Hospital, Basel, Switzerland (Unknown); Klinikum Kempten, Kempten, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12032024
Record Dates: First submitted 2024-03-28; First posted 2024-04-15 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Ventral Hernia; Incisional Hernia; Abdominal Wall Defect
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients are blinded to their treatment allocation until hospital discharge criteria according to the primary endpoint are fulfilled. After discharge, blinding is difficult to be ensured because there is no control, if dressing have been removed or modified. To ensure patient blinding during hospital stay, patients from both treatment arms will receive identical dressings as if an open and minimal-invasive access had been performed. In case the dressing must be changed during the hospital stay, this will be performed while the patient is blinded using a cover.
  In case for any reason the patient has been unblinded to his treatment allocation (accidental or intentional dressing removal, bed-side wound opening, other) all outcome data are assessed regardless and unblinding is documented and reported in the final report.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotically-assisted ventral hernia repair (RVHR) (Experimental)
  Interventions: Procedure: Robotically-assisted ventral hernia repair (RVHR)
- Open ventral hernia repair (OVHR) (Active Comparator)
  Interventions: Procedure: Open ventral hernia repair (OVHR)

INTERVENTIONS:
Procedure: Robotically-assisted ventral hernia repair (RVHR) — 3 8mm robotic trocars are placed intraabdominally and the DaVinci Xi-robotic system is docked. Adhesiolysis from any adherent structures to the abdominal wall is performed. Incision of the lateral verge of the retromuscular space and retromuscular dissection. Superior and inferior cross-over to the contralateral retromuscular space and dissection of the hernia sac.
  Unilateral or bilateral transversus abdominis release (TAR) is performed, if necessary. Running suture with absorbable barbed suture of the posterior rectus sheath and peritoneum, as appropriate. Synthetic retromuscular mesh placement with a mesh-size as large as the prepared surface allows. Closure of the anterior rectus sheath with absorbable barbed running suture. Port extraction, skin closure. Dressing from xyphoid to pubis and 6 lateral dressings for blinding purposes.
  Arms: Robotically-assisted ventral hernia repair (RVHR)
Procedure: Open ventral hernia repair (OVHR) — Median laparotomy with a minimal length of the previous scar (in case of incisional hernia) and adhesiolysis is performed, where necessary, to liberate the abdominal wall and the ventral hernia from adhesions. Bilateral dissection of the posterior rectus sheath under visualisation and sparing of the epigastric vessels and neurovascular bundles. Closure of the posterior rectus sheath with a slowly-absorbable running suture. Indication for a uni- or bilateral TAR identical to the intervention group. Retromuscular synthetic mesh placement with a mesh-size as far as the prepared surface allows. Mesh fixation optional with either absorbable sutures to the posterior sheath or with glubran glue. Closure of the anterior rectus sheath with a slowly-absorbable running suture. Skin closure. Dressing from xyphoid to pubis and 6 lateral dressings for blinding purposes.
  Arms: Open ventral hernia repair (OVHR)

SUMMARY:
This study investigates on the effect of two different operative techniques to treat large abdominal wall defects.

The goal of this clinical trial is to learn if the minimally-invasive, robotically-assisted ventral hernia repair (RVHR) leads to a better outcome than the open ventral hernia repair (OVHR).

The main questions it aims to answer are:

length of stay after the operation rate of complications rate of recurrence and reoperations quality of life.

Participants will:

Either be operated using the RVHR or OVHR will be followed up either in person or via email / phone call at day 7, day 30, 6 months, 1, 3 and 5 years after the surgery to asses the above-stated main and some more outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 years
* Informed consent obtained
* Transverse diameter of ventral hernia >4cm - 15cm
* Eligible to open and minimally-invasive surgery according to preoperative anaesthetic assessment

Exclusion Criteria:

* precedent hernia treatment with mesh placement in the retromuscular space
* precedent anterior or posterior component separation or transversus abdominis release (TAR)
* active wound infection
* current cancer diagnosis
* presence of ileostomy, colostomy or ileal conduit
* liver disease defined by the presence of ascites
* end-stage renal disease requiring dialysis
* need of an emergency surgery
* pregnancy

Criteria for participating surgeons Each participating surgeon has performed 20 or more OVHR and RVHR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: length of stay | 30 days
  Length of stay Length of stay is defined as the time from the operation until patient discharge is feasible according to the following criteria:
  * pain on numeric rating scale (NRS) < 4 without opioid use
  * tolerance of oral food intake without nausea / vomiting
  * no signs of surgical site occurrence (SSO) or other postoperative complications
  * no drains in place
  * autonomy in daily living activities

SECONDARY OUTCOMES:
Comprehensive complication index (CCI) | 30 days
  According to Slankamenac K, Graf R, Barkun J, Clavien P. The Comprehensive Complication Index. Ann Surg. 2013;258 The CCI ranges from 0 (no complications) to maximum 100 (death of the patient).
Adverse events | 30 days
  * Intraoperative adverse events (bleeding, conversion rate, injury to bowel structures)
  * Postoperative adverse events (all other than surgical site occurrences such as ileus, pulmonary embolism, pneumonia, etc.) according to Clavien-Dindo Classification up to 30 days after surgery.
pain after surgery | 5 years
  - Pain, measured using the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity Short Form 3a after 7days, 30 days, 6 months, 1, 3 and 5 years.
  The range fro the PROMIS ranges from 3 (no pain) to maximum of 15 (very severe pain) points.
Functional recovery | 5 years
  Functional recovery measured using the European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) Questionnaire.
  The questionnaire uses 5 questions describing the patients health and abilities on that particular day and a visual analogue scale question (0 = worst, 100 = best) on the patients health on that particular day.
Quality of life using SF-12 form | 5 years
  The 12-item Short Form Survey (SF-12) is a general health questionnaire that was first published in 1995 as part of the Medical Outcomes Study (MOS). The SF-12 was constructed using questions drawn from each of the 8 dimensions of the MOS 36 item Short Form Survey (SF-36).
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12).
  The score ranges from 0 - 100, with a higher score indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Baur, MD, Principal Investigator — Clarunis - Universitäres Bauchzentrum Basel; Julian Süsstrunk, MD, Principal Investigator — Clarunis - Universitäres Bauchzentrum Basel

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data (IPD) may be shared upon reasonable request. If IPD is shared, data will be anonymised completely.